CLINICAL TRIAL: NCT01943253
Title: Water-jet Assisted Endoscopic Submucosal Dissection (ESD) in Comparison to Conventional ESD Technique for Treatment of Early Gastric Cancer
Brief Title: Water-jet Assisted ESD vs Conventional ESD Technique for Treating Early Gastric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Evangelisches Krankenhaus Düsseldorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hybrid ESD
Record Dates: First submitted 2013-09-04; First posted 2013-09-16 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Stomach Neoplasms
Keywords: Early gastric cancer,; endoscopic submucosal dissection (ESD); water-jet assisted ESD
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional ESD (Active Comparator): Conventional ESD: Conventional ESD technique using IT2-Knife, Dual-Knife, Hook-Knife (Olympus Europe, Hamburg, Germany) ERBE VIO 300D (V2.1.4) RF-surgery system (ERBE Elektromedizin GmbH, Tübingen, Germany) Injection of fluid: Syringe
  Interventions: Device: Conventional ESD
- Hybridknife ESD (Active Comparator): Group 2: Water-jet assisted HybridKnife® ESD technique using HybridKnife® (Erbe Elektromedizin GmbH, Tübingen, Germany) ERBE VIO 300D (V2.1.4) RF-surgery system (ERBE Elektromedizin GmbH, Tübingen, Germany)
  Injection of fluid: Integrated in HybridKnife® with ERBEJet 2 water-jet surgery system (ERBE Elektromedizin GmbH, Tübingen, Germany)
  Interventions: Device: Hybridknife ESD

INTERVENTIONS:
Device: Conventional ESD — Conventional ESD: Conventional ESD technique using IT2-Knife, Dual-Knife, Hook-Knife (Olympus Europe, Hamburg, Germany; Olympus Japan) ERBE VIO 300D (V2.1.4) RF-surgery system (ERBE Elektromedizin GmbH, Tübingen, Germany) Injection of fluid: Syringe
  Arms: Conventional ESD
Device: Hybridknife ESD — Group 2: Water-jet assisted HybridKnife® ESD technique using HybridKnife® (Erbe Elektromedizin GmbH, Tübingen, Germany) ERBE VIO 300D (V2.1.4) RF-surgery system (ERBE Elektromedizin GmbH, Tübingen, Germany) Injection of fluid: Integrated in HybridKnife® with ERBEJet 2 water-jet surgery system (ERBE Elektromedizin GmbH, Tübingen, Germany)
  Other Names: Water-jet assisted HybridKnife® ESD
  Arms: Hybridknife ESD

SUMMARY:
1. Introduction The aim of the study is to evaluate the efficacy and safety of ESD by use of a new water-jet assisted ESD system using the HybridKnife® in patients with early gastric neoplastic lesions in comparison to the conventional ESD established in Japan. The water-assisted ESD technology allows pressure controlled injection of fluids through the tip of a recently developed HybridKnife®. Submucosal injection, circumferential cutting and dissection of lesions as well as coagulation of bleeding can be performed with the same device without need for changing the instrument. These options should accelerate the procedure and may increase its safety and efficacy.
2. Hypothesis The water-jet assisted ESD technique using the HybridKnife® bears the advantage of less instrument changes due to the combination of high-frequency cutting and water-jet application in one single instrument. This should lead to a simplified ESD procedure, shorter learn-ing curve and especially to a shorter procedure time.

The water-jet assisted ESD technique should be shorter than the conventional ESD techniques using IT2-, Dual- and Hook-Knifes at least with the same safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* adults (≥ 18 years) with confirmed diagnosis of gastric adenoma or early gastric adenocarcinoma
* differentiated mucosal adenocarinoma without ulcer findings ≤ 60 mm in diameter.
* Lesions with ulceration ≤ 30 mm in diameter.
* undifferentiated type of mucosal cancer is ≤ 20 mm.
* The patient has given written informed consent.

Exclusion Criteria:

* pregnancy
* coagulopathy (INR>2.0, platelets < 70/nl)
* mucosal lesions which did not meet the inclusion criteria
* evidence of local or distant metastases according to endoscopic ultrasound (EUS) and/or CT scan, EUS (7.5 MHz probe) findings of tumor infiltration into deep layers of the submucosa or muscularis propria. -Patients unfit for deep sedation by use of propofol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2011-05; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Procedure time | during procedure
  The primary objective of the study is the procedure time of ESD using the conventional ESD technique in comparison to the water-jet assisted HybridKnife®-ESD technique.

SECONDARY OUTCOMES:
en bloc resection rate | in procedure
  Resection of the targeted lesion including coagulation markers in one piece.
histological R0 rate | 7 days after procedure
  En-bloc resection and histological confirmation of horizontal and vertical free margins of neoplasia.
Histologically incomplete resection | 7 days after procedure
  Tumor infiltrated (R1) or undetermined (RX) margins of the resected specimen.
procedure related morbidity and mortality and complication rate | 30 days after procedure
  procedure related morbidity and mortality
complication rate | 30 days after procedure
  any complication occurs after procedure within 30 days, such as bleeding or perforation rates

CONTACTS AND LOCATIONS:
Overall Officials: Horst Neuhaus, Study Director — Evangelisches Krankenhaus Düsseldorf; Pinghong Zhou, Principal Investigator — Endoscopy Center, Zhongshan Hospital, Fudan University
Locations (1):
- Evangelisches Krankenhaus Düsseldorf, Düsseldorf, Germany